CLINICAL TRIAL: NCT06492499
Title: Patient-Centric Innovation: Superior Vena Cava Approach in Zero-Fluoroscopy Radiofrequency Catheter Ablation for Atrioventricular Nodal Reentrant Tachycardia
Brief Title: Patient-Centric Innovation: Superior Vena Cava Approach in Zero-Fluoroscopy
Status: Completed | Type: Observational
Sponsor: Ning Zhou (Other)
Responsible Party: Sponsor-Investigator, Ning Zhou, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: m202276475
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Atrioventricular Nodal Reentrant Tachycardia
Keywords: Zero-Fluoroscopy; Superior Vena Cava (SVC) Approach; Radiofrequency Catheter Ablation
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SVC Approach Group: This group includes patients who underwent zero-fluoroscopy radiofrequency catheter ablation (RFCA) for atrioventricular nodal reentrant tachycardia (AVNRT) using the superior vena cava (SVC) approach. The catheter was inserted through the median cubital vein or basilic vein, navigating through the axillary vein, subclavian vein, and brachiocephalic vein to reach the SVC. The ablation procedure was performed under conscious sedation and local infiltration anesthesia, with a large-tip electrode catheter used for mapping and ablation guided by the EnSite NavX system. The ablation parameters were set at 40 W power and 50°C temperature.
  Interventions: Procedure: Zero-Fluoroscopy Radiofrequency Catheter Ablation
- IVC Approach Group: This group includes patients who underwent zero-fluoroscopy radiofrequency catheter ablation (RFCA) for atrioventricular nodal reentrant tachycardia (AVNRT) using the inferior vena cava (IVC) approach. The catheter was inserted through the femoral vein, extending through the iliac vein to the IVC. The ablation procedure was performed under conscious sedation and local infiltration anesthesia, with a large-tip electrode catheter used for mapping and ablation guided by the EnSite NavX system. The ablation parameters were set at 40 W power and 50°C temperature.

INTERVENTIONS:
Procedure: Zero-Fluoroscopy Radiofrequency Catheter Ablation — Patients undergo zero-fluoroscopy RFCA for atrioventricular nodal reentrant tachycardia (AVNRT) using the superior vena cava (SVC) or inferior vena cava (IVC) approach. The procedure is performed under conscious sedation and local infiltration anesthesia. A large-tip electrode catheter is used for mapping and ablation, guided by the EnSite NavX system, with ablation parameters set at 40 W power and 50°C temperature.
  Groups: SVC Approach Group

SUMMARY:
This study aims to evaluate the viability and therapeutic efficacy of zero-fluoroscopy radiofrequency catheter ablation (RFCA) using the superior vena cava (SVC) approach in patients with atrioventricular nodal reentrant tachycardia (AVNRT). The study compares outcomes between the SVC approach and the conventional inferior vena cava (IVC) approach. Patients diagnosed with AVNRT who underwent RFCA between June 2022 and October 2022 were retrospectively analyzed. The primary outcome measure is the non-inducibility of AVNRT, while secondary outcomes include postoperative recovery time and complication rates. The study seeks to provide a safer and more efficient RFCA method, enhancing patient recovery by minimizing radiation exposure and optimizing catheter access routes.

DETAILED DESCRIPTION:
This retrospective study investigates the feasibility and therapeutic efficacy of zero-fluoroscopy radiofrequency catheter ablation (RFCA) using the superior vena cava (SVC) approach in patients diagnosed with atrioventricular nodal reentrant tachycardia (AVNRT). The study was conducted at our institution between June 2022 and October 2022, including adult patients (age >18 years) who underwent RFCA during this period. Patients were divided into two groups based on the catheter access site: the SVC approach group and the inferior vena cava (IVC) approach group.

The primary objective of the study is to assess the success rate of AVNRT ablation using the SVC approach compared to the conventional IVC approach, under zero-fluoroscopy conditions. Secondary objectives include evaluating the postoperative recovery time, incidence of complications, and overall patient outcomes.

Inclusion criteria required that patients experienced at least one episode of AVNRT during transesophageal atrial pacing (TEAP) and programmed stimulation. Exclusion criteria included cases where AVNRT was attributed to reversible causes such as acute myocarditis, cardiac surgery, or other types of tachycardias (e.g., atrial tachycardia, Wolff-Parkinson-White syndrome, ventricular tachycardia).

The electrophysiologic study involved TEAP and programmed stimulation to screen for AVNRT and exclude other arrhythmias. The catheterization procedure was performed under conscious sedation and local infiltration anesthesia, with continuous monitoring of vital signs. Catheter access sites for the SVC group included the median cubital vein and the basilic vein, while the femoral vein was used for the IVC group. The ablation procedure utilized a large-tip electrode catheter for mapping and ablation, guided by the EnSite NavX system.

Ablation endpoints were determined by the non-inducibility of AVNRT after programmed stimulation. Follow-up evaluations included monitoring for recurrence of atrial arrhythmias or the occurrence of iatrogenic atrioventricular block (AVB). Statistical analysis was performed using R 4.4.0 software, with continuous variables expressed as mean ± SD or median (interquartile range) and categorical variables as counts or percentages. An unpaired t-test or nonparametric test was used to compare the SVC and IVC approach groups, with a p-value of <0.05 considered statistically significant.

This study aims to demonstrate that the SVC approach for zero-fluoroscopy RFCA is a viable and effective alternative to the conventional IVC approach, potentially offering advantages such as reduced postoperative vascular events and elimination of bed rest requirements. The findings could broaden treatment options and enhance patient safety in RFCA procedures. Further research is encouraged to validate these findings across diverse populations and optimize procedural techniques for improved long-term efficacy and minimized risks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 years.
* Diagnosed with atrioventricular nodal reentrant tachycardia (AVNRT).
* Underwent radiofrequency catheter ablation (RFCA) at our institution between June 2022 and October 2022.
* Experienced at least one episode of AVNRT during transesophageal atrial pacing (TEAP) and programmed stimulation.
* Provided informed consent for the procedure and data collection.

Exclusion Criteria:

* AVNRT attributed to reversible causes, such as acute myocarditis or recent cardiac surgery.
* Presence of other types of tachycardias (e.g., atrial tachycardia, Wolff-Parkinson-White syndrome, ventricular tachycardia).
* Inability to abstain from pharmacological interventions for at least five half-lives of the medication prior to TEAP.
* Contraindications for the use of conscious sedation or local anesthesia.
* Severe comorbidities that would interfere with study participation or follow-up.
* Patients who are pregnant or lactating.
* Previous RFCA procedures for AVNRT within the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults (age >18 years) diagnosed with AVNRT who underwent RFCA at our institution between June and October 2022. Patients were divided into two groups based on catheter access site: the SVC approach group (median cubital or basilic vein) and the IVC approach group (femoral vein). Inclusion required at least one AVNRT episode during TEAP and programmed stimulation. Exclusion criteria were reversible causes of AVNRT, other tachycardias, severe comorbidities, or contraindications for conscious sedation or local anesthesia. This setup allows comparative analysis of SVC and IVC approaches focusing on success, complications, and recovery.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Non-inducibility of Atrioventricular Nodal Reentrant Tachycardia (AVNRT) | During the procedure
  This is determined during the procedure by performing programmed stimulation to test for the presence of AVNRT. Non-inducibility is confirmed if AVNRT cannot be induced following the ablation, indicating a successful therapeutic intervention.
Recurrence of supraventricular tachycardia | Within 1 year post-procedure
  It is defined as any documented episode of supraventricular tachycardia, such as AVNRT, atrial fibrillation, or atrial flutter, confirmed by electrocardiographic evidence.

SECONDARY OUTCOMES:
Postoperative Recovery Time | Within 24 hours post-procedure
  It is defined as the duration from the completion of the RFCA procedure to the patient's ability to walk unassisted.
Complication Rate | Within 1 year post-procedure
  It is defined as any documented episode of SVT, including AVNRT, confirmed by electrocardiographic evidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No